CLINICAL TRIAL: NCT01652014
Title: Hematopoietic Stem Cell Transplantation Using Alternate Donor Umbilical Cord Blood Options
Brief Title: Single or Double Donor Umbilical Cord Blood Transplant in Treating Patients With High-Risk Hematologic Malignancies
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 021002; NCI-2011-03187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0220100266 (Other: IRB Number); P30CA072720 (NIH)
Record Dates: First submitted 2012-07-20; First posted 2012-07-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Blastic Phase Chronic Myelogenous Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
Keywords: Transplantation; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Blast Crisis; Intraocular Lymphoma; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Transplantation; Whole-Body Irradiation; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Double UCB transplantation
  Patients receive conditioning comprising fludarabine phosphate IV over 30 minutes on days -6 to -2, cyclophosphamide IV over 1 hour on day -6, and undergo TBI on day -1. Patients also receive GVHD prophylaxis comprising tacrolimus IV continuously or PO beginning on day -3 with taper and mycophenolate mofetil PO BID days 1-30. Patients undergo double allogeneic UCB transplant on day 0.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: double-unit umbilical cord blood transplantation; Radiation: total-body irradiation; Drug: tacrolimus
- Arm II (Experimental): Sub-threshold single UCB + irradiated PBMCs transplantation
  Patients receive conditioning comprising fludarabine phosphate IV over 30 minutes on days -6 to -2, cyclophosphamide IV over 1 hour on day -6, and undergo TBI on day -1. Patients also receive GVHD prophylaxis comprising tacrolimus IV continuously or PO beginning on day -3 with taper and mycophenolate mofetil PO BID days 1-30. Patients undergo single allogeneic UCB transplant on day 0. Patients also undergo irradiated allogeneic PBMC transplant within 8 hours following the UCB infusion.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: total-body irradiation; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: cyclophosphamide — Given IV over 1 hour on Day -6; after pre-hydration
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: fludarabine phosphate — Given IV daily over 30 minutes for 5 days (Days -6 to -2)
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: mycophenolate mofetil — Given PO 1.0 g BID Day 1-30
  Other Names: Cellcept; MMF
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo double-unit allogeneic UCB transplant
  Arms: Arm I
Procedure: umbilical cord blood transplantation — Undergo single allogeneic UCB transplant
  Other Names: cord blood transplantation; transplantation, umbilical cord blood; UCB transplantation
  Arms: Arm II
Procedure: double-unit umbilical cord blood transplantation — Undergo double-unit allogeneic UCB transplant
  Arms: Arm I
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: tacrolimus — Given IV 0.03 mg/kg/d as continuous infusion over 24 hours starting Day -3 with dose adjustments to maintain level of 8-20 mg/ml
  Other Names: FK 506; Prograf
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo single allogeneic UCB transplant
  Arms: Arm II
Procedure: peripheral blood stem cell transplantation — Undergo irradiated allogeneic peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
  Arms: Arm II

SUMMARY:
This study will determine the safety and applicability of experimental forms of umbilical cord blood (UCB) transplantation for patients with high risk hematologic malignancies who might benefit from a hematopoietic stem cell transplant (HSCT) but who do not have a standard donor option (no available HLA-matched related donor (MRD), HLA-matched unrelated donor (MUD)), or single UCB unit with adequate cell number and HLA-match).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven hematologic malignancy with anticipated 2 year survival < 20% with standard therapy; patients age <18 are excluded by virtue of the policies and procedures of the allogeneic hematopoietic stem cell transplant (HSCT) program (Cancer Institute of New Jersey [CINJ]/Robert Wood Johnson University Hospital [RWJUH] is not an approved Pediatric Transplant Center); patients > age 65 are generally not considered candidates for experimental unrelated allogeneic HSCT, as utilized in this study by virtue of the anticipated delayed immune reconstitution, high risk of GVHD, and known negative impact of age on outcomes
* Patients eligible for this trial will have high risk diseases that include, but are not limited to:

  * Acute myeloid leukemia (AML) in second complete remission (CR2) or greater or early relapse with < 5% marrow blasts and no circulating blasts
  * AML in first complete remission (CR1) with high risk cytogenetics (complex, monosomy 5, monosomy 7, 11q23 (not t(9;11)), t(6;9), chromosome 3, monosomy phenotype and other karyotypes estimated to have =< 20% disease free survival at 3 years) or secondary/transformed AML without favorable cytogenetics;
  * Acute lymphoblastic leukemia (ALL) with t(9;22), 11q23 abnormality or early relapse (< 5% marrow blasts) or CR2 or greater;
  * Chronic myeloid leukemia (CML) resistant/refractory to all commercially available Abelson (abl) kinase inhibitors (e.g. imatinib mesylate, dasatinib, nilotinib) or predicted to be so based upon clinical course or abl kinase domain mutation analysis; or in accelerated phase or blast crisis;
  * High intermediate to high international prognostic score myelodysplasia;
  * Non-Hodgkin lymphoma (NHL)/Hodgkin lymphoma (HL)/other lymphoproliferative diseases resistant/refractory to standard therapies and for whom an autologous transplant is considered to be inappropriate (e.g. bone marrow involvement, chemotherapy refractory disease, prior transplant);
  * Chronic lymphocytic leukemia (CLL) resistant/refractory to standard therapies (e.g. fludarabine) or high risk cytogenetics/fluorescence in situ hybridization (FISH) (e.g. 17p-);
  * Myeloproliferative disorders with progressive disease or cytopenias or clinical symptoms refractory to standard therapy (e.g. hypomethylating agents)
  * Relapsed or refractory multiple myeloma after (or not eligible for) high dose chemotherapy/autologous hematopoietic stem cell rescue and following salvage therapy with thalidomide, lenalidomide or bortezomib/other Food and Drug Administration (FDA)-approved multiple myeloma salvage therapies;
  * Other hematologic malignancies/disorders with anticipated 2 year survival < 20%, as established by available data bases, medical literature and the documented consensus of the Hematologic Malignancies Tumor Study Group
* Patients must be an allogeneic HSCT candidate but have no standard donor (matched related donor [MRD], human leukocyte antigen [HLA]-matched unrelated donor [MUD] or single UCB unit of appropriate size and HLA type) available
* Patients must have available UCB unit(s)
* Patients considered for Arm 2 must not be eligible for Arm 1 and must have an HLA-haploidentical sibling, parent, child, or other relative (uncle, aunt, first cousin, niece or nephew) who meets donor requirements as outlined in Donor Eligibility criteria
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Left ventricular (LV) ejection fraction >= 50%
* Diffusion capacity of carbon monoxide (DLCO) corrected for hemoglobin > 60%
* Total bilirubin within normal institutional limits unless the patient has Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (ULN)
* Measured or estimated creatinine clearance > 50 ml/min
* Hematopoietic stem cell co-morbidity index =< 2
* There must be a negative pregnancy test for women of childbearing potential within 1 week of therapy; there must be willingness to avoid pregnancy and undergo counseling about contraceptive techniques throughout the course of treatment
* There must be no uncontrolled infections or active acute or chronic illnesses such as diabetes, angina/myocardial ischemia, cardiac arrhythmia, venous thrombosis/embolism, cerebrovascular disease, seizure disorder, psychiatric illness or other intercurrent illness that is not well controlled or is anticipated to be difficult to control during the proposed therapy
* The patient must be aware of the high risk and experimental nature of the treatment and provide informed consent
* The patient must have clearance for HSCT after psychosocial evaluation
* The patient must have adequate insurance or other support to meet the anticipated financial burden imposed by the costs of therapy
* DONOR (for allogeneic lymphocytes, Arm 2 only): Relative (parent, child, sibling, first cousin, uncle aunt, nephew, niece) with appropriate HLA match (>= 3/6 HLA A, B, DR match)
* DONOR (for allogeneic lymphocytes, Arm 2 only): Age >= 18 years old
* DONOR (for allogeneic lymphocytes, Arm 2 only): Normal hemogram; potential donors not having a normal hemogram may be utilized at the discretion of the Principal Investigator
* DONOR (for allogeneic lymphocytes, Arm 2 only): Not pregnant or lactating
* DONOR (for allogeneic lymphocytes, Arm 2 only): Not human immunodeficiency virus (HIV)-1, HIV-2, hepatitis C (HCV), Hepatitis B core or human T-lymphotropic virus (HTLV)-I/II seropositive; hepatitis B surface antigen (HB Sag)(-); must meet other infectious disease screening criteria utilized by New Brunswick Affiliated Hospital (NBAH) Blood Center
* DONOR (for allogeneic lymphocytes, Arm 2 only): No uncontrolled infections, other medical or psychological/social conditions, or required medications that might increase the likelihood of patient or donor adverse effects or poor outcomes
* DONOR (for allogeneic lymphocytes, Arm 2 only): Meet other blood bank criteria for blood product donation (as determined by NBAH Blood Center screening history)
* DONOR (for allogeneic lymphocytes, Arm 2 only): Donors must be informed of the investigational nature of this study, understand the requirements, potential benefits and potential risks of the experimental treatment, and give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Prior extensive radiation therapy that the radiation oncologist feels precludes additional TBI
* Patients with known human immunodeficiency virus (HIV) are excluded due to side effects of the therapy on the immune system
* Patients with known active central nervous system (CNS) disease will be excluded from this clinical trial because they often develop progressive neurologic dysfunction unresponsive to HSCT therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Engraftment of white blood cells (WBC) (absolute neutrophil count > 500/mm^3) | 3 years
Non-relapse mortality | 40 months

SECONDARY OUTCOMES:
Platelet engraftment rate (non-transfusion dependent) | At 100 days
Transplant related mortality | At 1 year
Rates of infection requiring hospitalization or prolongation of hospitalization | Up to 2 years
Incidence of steroid-refractory acute GVHD | at 100 days
  GVHD will be staged per standard guidelines of the American Society for Blood and Bone Marrow Transplantation.
Incidence of extensive chronic GVHD | up to 2 years
  GVHD will be staged per standard guidelines of the American Society for Blood and Bone Marrow Transplantation.
Total time on immunosuppressive therapy | Up to 2 years
Time to CD4 count > 200/mm^3 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States